CLINICAL TRIAL: NCT00344968
Title: A Randomized, Double-Masked, Parallel Group, Multi-center, Dose-Finding Comparison of the Safety and Efficacy of ASI-001A 0.5 μg/Day and ASI-001B 0.2 μg/Day Fluocinolone Acetonide Intravitreal Inserts to Sham Injection in Subjects With Diabetic Macular Edema
Brief Title: Fluocinolone Acetonide Implant Compared to Sham Injection in Patients With Diabetic Macular Edema
Acronym: FAME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-01-05-001
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: fluocinolone acetonide
- 2 (Experimental)
  Interventions: Drug: Fluocinolone Acetonide
- 3 (Sham Comparator)
  Interventions: Procedure: Standard of care laser photocoagulation

INTERVENTIONS:
Drug: fluocinolone acetonide — 0.5 mg fluocinolone acetonide intravitreal insert
  Arms: 1
Drug: Fluocinolone Acetonide — 0.2 mg fluocinolone acetonide intravitreal insert
  Arms: 2
Procedure: Standard of care laser photocoagulation — Laser photocoagulation
  Arms: 3

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal insert of fluocinolone acetonide for the treatment of diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years with diabetic macular edema
* Diagnosis of diabetes mellitus types 1 or 2
* Best corrected visual acuity of 19-68 letters
* Retinal thickness > 250 micron by OCT
* Investigator is comfortable deferring macular laser treatment for 6 weeks

Exclusion Criteria:

* Glaucoma, ocular hypertension, IOP >21 mmHg or concurrent therapy at screening with IOP lowering agents
* Retinal or choroidal neovascularization due to ocular conditions other than diabetic retinopathy
* Prior intravitreal, subtenon, or periocular steroid therapy within 6 months
* Any ocular surgery within the last 3 months
* Retinal laser treatment within the last 3 months
* History of uncontrolled IOP elevation with steroid use that did not respond to topical therapy
* Any lens opacity which impairs visualization of the posterior pole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 956 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta, Georgia, United States

REFERENCES:
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Holden SE, Kapik B, Beiderbeck AB, Currie CJ. Comparison of data characterizing the clinical effectiveness of the fluocinolone intravitreal implant (ILUVIEN) in patients with diabetic macular edema from the real world, non-interventional ICE-UK study and the FAME randomized controlled trials. Curr Med Res Opin. 2019 Jul;35(7):1165-1176. doi: 10.1080/03007995.2018.1560779. Epub 2019 Jan 17. PMID 30569759

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Comparator: Procedure: Standard of care laser photocoagulation
- Fluocinolone Acetonide: 0.2 ug/Day Implant: Dose 0.2 ug/day Medidur Implant
- Fluocinolone Acetonide: 0.5 ug/Day Implant: Dose 0.5 ug/day Medidur implant
Period: Overall Study
Arm/Group | Sham Comparator | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Started | 185 | 376 | 395
Completed | 126 | 274 | 279
Not Completed | 59 | 102 | 116
Not completed — Adverse Event | 5 | 4 | 15
Not completed — Unsatisfactory Therapeutic Effect | 3 | 0 | 1
Not completed — Protocol Violation | 2 | 2 | 5
Not completed — Withdrawal by Subject | 14 | 31 | 27
Not completed — Lost to Follow-up | 24 | 37 | 37
Not completed — Death | 11 | 27 | 31
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Three subjects were randomized but did not receive treatment. These subjects were not included in the safety analysis, which accounts for the discrepancy in the overall number of participants.
Groups:
- 0.2 ug/Day Implant: Dose 0.2 ug/day Medidur Implant
- 0.5 ug/Day Implant: Dose 0.5 ug/day Medidur implant
- Total: Total of all reporting groups
Arm/Group | Sham Comparator | 0.2 ug/Day Implant | 0.5 ug/Day Implant | Total
Number analyzed (Participants) | 185 | 376 | 395 | 956
Age, Categorical [Number; unit: participants] — Three subjects were randomized but did not receive treatment. These subjects were not included in the safety analysis, which accounts for the discrepancy in the overall number of participants.
  participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 119 | 213 | 232 | 564
    >=65 years | 66 | 162 | 161 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] — Three subjects were randomized but did not receive treatment. These subjects were not included in the safety analysis, which accounts for the discrepancy in the overall number of participants.
  years | 61.9 (9.6) | 63.0 (9.3) | 62.2 (9.3) | 62.5 (9.4)
Gender [Number; unit: participants] — Three subjects were randomized but did not receive treatment. These subjects were not included in the safety analysis, which accounts for the discrepancy in the overall number of participants.
  participants
    Female | 77 | 160 | 150 | 387
    Male | 108 | 215 | 243 | 566
Region of Enrollment [Number; unit: participants] — Three subjects were randomized but did not receive treatment. These subjects were not included in the safety analysis, which accounts for the discrepancy in the overall number of participants.
  participants
    North America | 129 | 259 | 274 | 662
    India | 39 | 80 | 82 | 201
    Europe | 17 | 37 | 39 | 93

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: The percentage of subjects with an increase from baseline of 15 or more letters in best corrected visual acuity letter score as assessed by ETDRS eye chart (study eye).
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Sham Comparator | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 185 | 376 | 395
percentage of subjects | 18.9 (18.01) | 28.7 (19.04) [-2.5 to -17.1] | 27.8 (18.96) [-1.8 to -16.1]

2. Secondary Outcome: Retinal Thickness
Description: Retinal images where sent to a reading center for analysis. Some images were not clear/distorted and could not be properly analyzed. This accounts for the discrepancy in the number of participants analyzed.
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Sham Comparator | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 182 | 369 | 388
microns | 146.1 (192.10) | 113.5 (151.46) | 131.8 (162.46)

ADVERSE EVENTS:
Description: Three subjects were randomized but did not receive treatment. These subjects were not included in the safety analysis, which accounts for the discrepancy in the overall number of participants.
Groups:
- Sham Comparator: Standard of care laser photocoagulation
Arm/Group | Sham Comparator | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Serious Adverse Events (participants affected / at risk) | 112/185 | 292/375 | 331/393
Other Adverse Events (participants affected / at risk) | 174/185 | 360/375 | 388/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Comparator (N=185) | Fluocinolone Acetonide: 0.2 ug/Day Implant (N=375) | Fluocinolone Acetonide: 0.5 ug/Day Implant (N=393)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 5 (9) | 6 (6)
Angina unstable (Cardiac disorders) | 0 (0) | 4 (5) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Bundle branch block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 4 (4) | 4 (4)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 8 (8) | 12 (17) | 16 (25)
Cardiac fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (5) | 10 (13) | 15 (15)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 14 (17) | 16 (17)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 2 (2) — #Study eye
Anterior capsule contraction (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Study eye
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Fellow eye
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Conjunctival ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Corneal thinning (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Diabetic retinal oedema (Eye disorders) | 1 (2) | 0 (0) | 0 (0) — #Study eye
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Fellow eye
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 1 (1) — #Study eye
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Study eye
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Fellow eye
Glaucoma (Eye disorders) | 2 (2) | 12 (12) | 12 (12) — #Study eye
Glaucoma (Eye disorders) | 1 (1) | 1 (1) | 3 (3) — #Fellow eye
Hyphaema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Hypotony of eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Iris adhesions (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Iris bombe (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Iris incarceration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Macular hole (Eye disorders) | 0 (0) | 2 (2) | 0 (0) — #Study eye
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Study eye
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Fellow eye
Maculopathy (Eye disorders) | 2 (5) | 2 (2) | 2 (2) — #Study eye
Maculopathy (Eye disorders) | 1 (1) | 1 (1) | 2 (2) — #Fellow eye
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 2 (2) — #Study eye
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 2 (2) — #Study eye
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Posterior capsule rupture (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Retinal artery embolism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Retinal detachment (Eye disorders) | 3 (4) | 2 (2) | 4 (4) — #Study eye
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 1 (1) — #Fellow eye
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Fellow eye
Scleral thinning (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 2 (2) — #Fellow eye
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Vitreous haemorrhage (Eye disorders) | 6 (8) | 10 (13) | 8 (9) — #Study eye
Vitreous haemorrhage (Eye disorders) | 8 (9) | 5 (6) | 9 (10) — #Fellow eye
Vitritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Study eye
Vitritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — #Fellow eye
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneum cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 8 (9) | 4 (4)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Polyp (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Blister infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 4 (6) | 6 (7)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) — #Study eye
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — #Fellow eye
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Gangrene (Infections and infestations) | 1 (1) | 1 (1) | 6 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (4) | 5 (7) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 13 (13) | 10 (12)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 5 (5)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tracheostomy infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — #Fellow eye
Chemical eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Eye operation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0) | 4 (4)
Diagnostic procedure (Investigations) | 0 (0) | 1 (2) | 0 (0)
Full blood count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hysteroscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 12 (16) | 20 (22) — #Study eye
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 2 (2) — #Fellow eye
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 3 (3)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 9 (12) | 10 (10)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 4 (5)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 5 (5)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 11 (13) | 10 (10)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (6) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 1 (2) | 4 (5) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Amputation revision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ankle operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 0 (0) | 2 (4) | 0 (0)
Arteriovenous graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bladder operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Blepharoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Blepharoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — #Fellow eye
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Carotid artery stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 33 (33) | 188 (188) | 231 (231) — #Study eye
Cataract operation (Surgical and medical procedures) | 32 (32) | 85 (85) | 87 (87) — #Fellow eye
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Colon operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
Cryotherapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — #Fellow eye
Dialysis device insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Eye excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — #Fellow eye
Eye operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — #Study eye
Foot operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Gallbladder operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Glaucoma surgery (Surgical and medical procedures) | 1 (1) | 7 (7) | 8 (10) — #Study eye
Glaucoma surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 5 (5) — #Fellow eye
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 3 (3)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intraocular lens extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2) — #Study eye
Iridotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1)
Pancreas transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Penile prosthesis insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ptosis repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Removal of foreign body from eye (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — #Study eye
Renal transplant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Retinal operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2) — #Study eye
Retinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) — #Fellow eye
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 4 (4) | 2 (2)
Trabeculectomy (Surgical and medical procedures) | 0 (0) | 10 (10) | 22 (22) — #Study eye
Trabeculoplasty (Surgical and medical procedures) | 0 (0) | 3 (5) | 10 (11) — #Study eye
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Uterine polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Vascular cauterisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 16 (16) | 19 (21) | 23 (30) — #Study eye
Vitrectomy (Surgical and medical procedures) | 13 (13) | 25 (27) | 27 (29) — #Fellow eye
Wound closure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — #Study eye
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arteritis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 3 (5) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Comparator (N=185) | Fluocinolone Acetonide: 0.2 ug/Day Implant (N=375) | Fluocinolone Acetonide: 0.5 ug/Day Implant (N=393)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 33 (36) | 42 (46)
Cataract (Eye disorders) | 53 (54) | 171 (183) | 213 (234) — #Study eye
Cataract (Eye disorders) | 46 (47) | 109 (115) | 121 (127) — #Fellow eye
Cataract subcapsular (Eye disorders) | 8 (9) | 28 (34) | 24 (34) — #Study eye
Conjunctival haemorrhage (Eye disorders) | 20 (21) | 43 (50) | 50 (62) — #Study eye
Dry eye (Eye disorders) | 11 (11) | 23 (24) | 22 (24) — #Study eye
Dry eye (Eye disorders) | 9 (9) | 23 (24) | 17 (18) — #Fellow eye
Eye irritation (Eye disorders) | 9 (11) | 27 (30) | 22 (22) — #Study eye
Eye pain (Eye disorders) | 22 (25) | 51 (57) | 65 (77) — #Study eye
Eye pain (Eye disorders) | 11 (11) | 17 (19) | 11 (11) — #Fellow eye
Maculopathy (Eye disorders) | 16 (21) | 22 (24) | 33 (36) — #Study eye
Maculopathy (Eye disorders) | 9 (9) | 16 (16) | 22 (25) — #Fellow eye
Myodesopsia (Eye disorders) | 13 (17) | 67 (80) | 68 (79) — #Study eye
Myodesopsia (Eye disorders) | 11 (12) | 17 (19) | 18 (19) — #Fellow eye
Posterior capsule opacification (Eye disorders) | 6 (6) | 32 (35) | 25 (27) — #Study eye
Posterior capsule opacification (Eye disorders) | 4 (4) | 19 (21) | 20 (20) — #Fellow eye
Retinal haemorrhage (Eye disorders) | 11 (13) | 9 (10) | 17 (18) — #Study eye
Vision blurred (Eye disorders) | 13 (16) | 28 (31) | 20 (22) — #Study eye
Vision blurred (Eye disorders) | 4 (5) | 21 (24) | 14 (15) — #Fellow eye
Visual acuity reduced (Eye disorders) | 17 (22) | 39 (44) | 35 (42) — #Study eye
Visual acuity reduced (Eye disorders) | 14 (19) | 25 (27) | 23 (35) — #Fellow eye
Visual impairment (Eye disorders) | 7 (8) | 13 (13) | 31 (35) — #Study eye
Vitreous detachment (Eye disorders) | 12 (12) | 26 (26) | 20 (20) — #Study eye
Vitreous haemorrhage (Eye disorders) | 25 (33) | 38 (52) | 46 (62) — #Study eye
Vitreous haemorrhage (Eye disorders) | 22 (32) | 36 (53) | 49 (65) — #Fellow eye
Constipation (Gastrointestinal disorders) | 7 (7) | 18 (20) | 27 (29)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (13) | 22 (22) | 26 (26)
Nausea (Gastrointestinal disorders) | 18 (21) | 28 (37) | 30 (32)
Vomiting (Gastrointestinal disorders) | 13 (14) | 15 (16) | 9 (11)
Nasopharyngitis (Infections and infestations) | 12 (17) | 22 (22) | 24 (26)
Sinusitis (Infections and infestations) | 7 (10) | 16 (17) | 22 (27)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 9 (10) | 20 (26)
Urinary tract infection (Infections and infestations) | 11 (14) | 20 (24) | 22 (26)
Intraocular pressure increased (Investigations) | 21 (22) | 129 (176) | 169 (244) — #Study eye
Intraocular pressure increased (Investigations) | 22 (22) | 40 (48) | 50 (67) — #Fellow eye
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 (13) | 24 (24) | 24 (24)
Headache (Nervous system disorders) | 10 (11) | 31 (33) | 21 (25)
Depression (Psychiatric disorders) | 7 (8) | 11 (12) | 22 (23)
Renal failure (Renal and urinary disorders) | 7 (7) | 19 (19) | 25 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 17 (17) | 21 (26)
Hypertension (Vascular disorders) | 29 (33) | 43 (50) | 57 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days